CLINICAL TRIAL: NCT00163007
Title: Nutritional Therapy for Patients With Acute Stroke and With Poor Nutritional Status or at Risk of Poor Nutritional Status
Brief Title: Nutritional Therapy for Stroke Patients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ostfold Hospital Trust (Other)
Collaborators: University of Oslo (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 297
Record Dates: First submitted 2005-09-09; First posted 2005-09-13 (Estimated); Last update posted 2009-05-11 (Estimated); Status verified 2009-05

CONDITIONS: Stroke; Malnutrition; Weight Loss; Dysphagia
MeSH Terms: conditions — Stroke; Malnutrition; Weight Loss; Deglutition Disorders | interventions — Nutritional Support

INTERVENTIONS:
Procedure: Nutritional support

SUMMARY:
Prospective, short-term studies in patients admitted for acute stroke have shown an increased risk of infections, bedsores, impaired functional outcome, slower rate of recovery, poorer rehabilitation potential and higher mortality in patients with a poor nutritional status. In hospitals without routine nutritional assessment and individual nutrition management plans, the risk of patients developing malnutrition may be increased. In this study, patients admitted for acute stroke are randomised into either receiving nutritional therapy derived from estimated individual nutritional intake and nutritional needs, or nutritional therapy based on routine care without routine assessment of nutritional status, intake, or needs. The primary outcome measure is the percentage of patients with weight loss ≥ 5 % at three month follow-up.

DETAILED DESCRIPTION:
Prospective, short-term studies in patients admitted for acute stroke have shown an increased risk of infections, bedsores, impaired functional outcome, slower rate of recovery, poorer rehabilitation potential and higher mortality in patients with a poor nutritional status. Sixteen percent of stroke patients are already malnourished on admission to hospital. The incidence of dysphagia in patients with acute stroke ranges from 30 to 45%. Dysphagia increases the risk of developing poor nutritional status, and new cases of malnutrition develop during the hospital stay, even during the first week. In hospitals without routine nutritional assessment and individual nutrition management plans, the risk of patients developing malnutrition may be increased. In this study patients admitted for acute stroke are randomised into either receiving nutritional therapy derived from estimated individual nutritional intake and nutritional needs, or nutritional therapy based on routine care; without routine assessment of nutritional status, intake or needs. Nutritional therapy: enriched meals, sip-feedings or enteral feedings. Parameters of nutritional status: Weight, BMI, TSF thickness, mid upper arm circumference, body composition, s-albumin and s-transferrin. Estimation of nutritional intake: Daily registration of food and drink intake. Estimating functional status: Hand grip strength, Barthels ADL index and Scandinavian stroke scale. Estimating quality of life: EQ-5D.

Before the inclusion started we decided to use the percentage of patients with weight loss ≥ 5 % at 3 months follow-up as the primary outcome measure because this is correlated better to clinical outcomes as e.g. mortality and comorbidity. Secondary outcome measures were then defined as handgrip strength, quality of life, nutritional status, nutrient intake and length of hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* Acute stroke based on clinical symptoms
* 18 years old and above
* < 7 days since debut of stroke symptoms and either body mass index (BMI) = or < 20
* Weight loss > 5% in 3-6 months or there has been little or is likely to be no or very little nutritional intake for > 5 days

Exclusion Criteria:

* Subarachnoidal bleeding and planned operation
* Severe dementia
* Reduced consciousness
* Immobility
* Expected short-time survival

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2005-05; Primary Completion 2008-03 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with weight loss >=5 % at three month follow-up.

SECONDARY OUTCOMES:
Quality of life, handgrip strength and nutritional status at three months. Dietary intake in hospital. Length of hospital stay.

CONTACTS AND LOCATIONS:
Overall Officials: Truls Hauge, PhD, Study Chair — Ullevaal University Hospital
Locations (1):
- Ostfold Hospital Trust, Fredrikstad, Norway

REFERENCES:
- [Derived] Ha L, Hauge T, Iversen PO. Body composition in older acute stroke patients after treatment with individualized, nutritional supplementation while in hospital. BMC Geriatr. 2010 Oct 18;10:75. doi: 10.1186/1471-2318-10-75. PMID 20955603
- [Derived] Ha L, Hauge T, Spenning AB, Iversen PO. Individual, nutritional support prevents undernutrition, increases muscle strength and improves QoL among elderly at nutritional risk hospitalized for acute stroke: a randomized, controlled trial. Clin Nutr. 2010 Oct;29(5):567-73. doi: 10.1016/j.clnu.2010.01.011. Epub 2010 Feb 21. PMID 20176418